CLINICAL TRIAL: NCT00876265
Title: A Randomized, Blinded, Controlled, Multicenter Study of the Safety and Effectiveness of Dermal Filler, Belotero®, After Mid-to-Deep Dermal Implantation for Correction of Moderate to Severe Facial Wrinkles
Brief Title: Multicenter Study of the Safety and Effectiveness of Dermal Filler, Belotero®.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MUS 90028-0622/1
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Facial Wrinkles
Keywords: Facial wrinkles; Nasolabial fold

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Belotero (Experimental)
  Interventions: Device: Belotero
- Zyplast (Active Comparator)
  Interventions: Device: Zyplast

INTERVENTIONS:
Device: Belotero — Belotero, injectable hyaluronic acid gel device, implanted into the nasolabial fold in the Treatment Phase of the study (multiple injections of 0.1 to 0.2 mL, up to a maximum of 3 mL over 2 treatment sessions). Dose was based on the severity of the wrinkle, with a maximum dose to achieve 100% correction to be administered.
  Arms: Belotero
Device: Zyplast — Zyplast Collagen Implant, an injectable dermal collagen device, implanted into the nasolabial fold in the Treatment Phase of the study (average injection of 1.0 mL). Dose was based on the severity of the wrinkle, with a maximum dose to achieve 100% correction to be administered. Zyplast was obtained by each site from commercially available supplies.
  Arms: Zyplast

SUMMARY:
This was a study to find out how an investigational product, Belotero, compares to a second product in people with facial wrinkles, such as nasolabial folds. Nasolabial folds are wrinkles on the face that go from the outside of the nostrils to the edges of the mouth. Additionally, this study determined Belotero is safe and tolerable and corrects facial wrinkles, such as nasolabial folds.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects reviewed and signed a statement of Informed Consent and a HIPAA authorization prior to initiating any study-specific procedures. In addition, subjects were asked to provide a separate release for use of their photographs in publications. Subjects could refuse the photo release without jeopardizing their eligibility to participate in the study.
2. Subjects were 18 - 75 years of age, and of any race or sex.
3. Female subjects were postmenopausal for at least 1 year, had a hysterectomy, or had a tubal ligation; or, if of childbearing potential, agreed to use an approved method of birth control throughout the study (i.e., oral/systemic contraceptives, intrauterine device [IUD], or spermicide in combination with a barrier method of contraception), were abstinent, or were in a monogamous relationship with a vasectomized partner; and had a negative urine pregnancy test at the screening visit.
4. Subjects had bilateral nasolabial folds with a severity score of 2 or 3 on the wrinkle SRS assessed by the blinded evaluator.
5. Each subject had an adequate understanding of the language (spoken and written English or Spanish) and was willing to comply with the study requirements.

Exclusion Criteria:

1. A personal history of allergic/anaphylactic reactions including hypersensitivity to local anesthetics (eg, lidocaine, etc), HA preparations, and/or gram-positive bacterial protein.
2. A known history of keloids or bleeding disorders.
3. An active inflammatory process in the nasolabial fold area (skin eruptions such as cysts, pimples, rashes, cancerous/pre-cancerous lesions, psoriasis, neurodermatitis, or any other active skin disease) or severe scarring that might interfere with study assessments.
4. Women who were pregnant, planning to become pregnant during the study, or who were breast-feeding.
5. Subjects who planned to undergo major facial surgery during the course of the study (eg, rhinoplasty [with or without implant], facelift, congenital defect repair, etc).
6. Subjects with clinically important disease, as judged by the investigator, within 3 months of the study (eg, significant laboratory test abnormalities, myocardial infarct, stroke, cancer, connective tissue diseases [scleroderma, systemic lupus erythematous], systemic infection, uncontrolled diabetes, etc.), including those with medical conditions that might require the use of immunosuppressive medications during the trial (eg, severe, uncontrolled asthma, rheumatoid arthritis, autoimmune diseases, etc).
7. Severe physical, neurological or mental disease.
8. Excessive facial hair that might interfere with the evaluation of the wrinkle assessments.
9. Any systemic or dermatologic disorder, which, in the opinion of the investigator,would interfere with the study results or increase the risk of adverse events (AEs).
10. Subjects who had used exclusionary medications/treatments.
11. Participation in a clinical investigation within the 30 days prior to the first planned device administration or during this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2006-12; Primary Completion 2007-07 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhoda Narins, MD, Principal Investigator — Dermatology Surgery and Laser Center
Locations (6):
- United States (6):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - Skin Care & Laser Physicians of Beverly Hills, Los Angeles, California
  - Maas Clinic, San Francisco, California
  - Savin Dermatology, New Haven, Connecticut
  - William Coleman, III, MD, Metairie, Louisiana
  - Dermatology Surgery and Laser Center, White Plains, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects in this trial were enrolled from six study centers in the United States between November 2006 and July 2007. Subjects were males or non-pregnant females aged 18 to 75 years and who had bilateral nasolabial folds with a severity of 2 or 3 (moderate to severe).
Pre-assignment Details: The planned enrollment was 120 subjects; 118 subjects were randomized.
Period: Overall Study
Arm/Group | Overall Study
Started | 118
Completed | 106
Not Completed | 12
Not completed — Miscellaneous reasons | 4
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 110
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 52.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Adjusted (LS) Mean Change From Baseline in Wrinkle Severity Rating Scale (SRS) Score of Each Nasolabial Fold (NLF) as Determined by the Blinded Evaluator at Week 12.
Description: The severity of the nasolabial folds was measured using the wrinkle Severity Rating Scale (SRS), where 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Extreme, which is an ordinal scale.
Time Frame: Baseline and Week 12 of follow-up
Population: The Full Analysis Set (FAS) population was the analysis population which was defined as all subjects who were randomized and received at least one injection of the study device to the nasolabial folds.
Measure: Least Squares Mean (Standard Error); unit: Wrinkle Severity Rating Score (SRS)
Groups:
- Belotero: Belotero was injected into the left or right nasolabial fold using a randomization schedule.
- Zyplast: Zyplast was injected into the opposite nasolabial fold that Belotero was injected into.
Arm/Group | Belotero | Zyplast
Number analyzed (Participants) | 118 | 118
Wrinkle Severity Rating Score (SRS) | 1.224 (0.111) [-0.228 to 0.323] | 1.176 (0.111)
Statistical Analysis 1: Comparison: Belotero vs Zyplast; The null, H0, and the alternative hypothesis, H1, are as follows: H0(1): adjusted mean(dadj[i]) ≤ -Δ versus H1(1): adjusted mean(dadj[i]) > -Δ H0(2): adjusted mean(dadj[i]) ≤ 0 versus H1(2): adjusted mean(dadj[i]) > 0 The sample size calculation was based on the following assumptions: Type I error α = 0.025 (one sided); Power = 90%; Non-inferiority margin Δ = 0.25; Estimated common standard deviation (SD) = 0.75. Under these assumptions, a total of 100 evaluable subjects were needed; Test type: Non-Inferiority or Equivalence — If the 95% CI or the difference between LS mean (Belotero) and LS mean (Zyplast) lies entirely above -Δ, noninferiority of Belotero will be concluded (first step). If, in addition, the CI lies entirely above 0, superiority of Belotero over Zyplast will be concluded (second step); p = 0.733, ANCOVA — Treatment term and all significant (p ≤ 0.10) covariate and covariate by treatment interactions will be retained in the final ANCOVA model. From the final ANCOVA model, adjusted (LS) means for Belotero and Zyplast was computed; Adjusted (LS) mean difference = 0.048, 95% CI 2-sided [-0.228 to 0.323], Standard Error of Mean 0.139

ADVERSE EVENTS:
Arm/Group | Belotero | Zyplast
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/118
Other Adverse Events (participants affected / at risk) | 108/118 | 109/118
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belotero (N=118) | Zyplast (N=118)
Injection site erythema (General disorders) | 67 | 75
Injection site swelling (General disorders) | 59 | 61
Injection site bruising (General disorders) | 66 | 51
Injection site pain (General disorders) | 49 | 58
Injection site discoloration (General disorders) | 28 | 31
Injection site pruritus (General disorders) | 16 | 24
Injection site induration (General disorders) | 10 | 14
Injection site nodule (Gastrointestinal disorders) | 8 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any proposed press release, announcement, disclosure for publication, whether or not in writing, prepared by or on behalf of Consultant as part of services under this Agreement or that relates to the work performed hereunder must be reviewed and approved in writing by Merz prior to dissemination.